CLINICAL TRIAL: NCT04464018
Title: The Effect of Hybrid Simulation in the Development of Intramuscular Injection Skills of Nursing Students
Brief Title: Nurse,Intramuscular Injection, Hybrid Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Arife Şanlıalp Zeyrek, prelector, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 60116787-020/4308
Record Dates: First submitted 2020-07-04; First posted 2020-07-09 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-07

CONDITIONS: Educational Problems
Keywords: intramuscular injection; hybrid simulation

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working group (Experimental): Working group (hybrid simulation method) after the theoretical lecture, the application with hybrid simulation method is made by videotaping. Repeat the same practice after 1 Week
  Interventions: Other: working grup
- Control group (No Intervention): Control group (Low reality simulation method) after the theoretical lecture, the application with low reality simulation method is made. Repeat the same practice after 1 Week Control group received only general care

INTERVENTIONS:
Other: working grup — After each student received theoretical training, they performed an intravenous injection on the model. In the study group performed hybrid simulation. After finishing the simulation application. the students went to the analysis room and watched their own application videos. The analysis session was held immediately after all the students in the group completed their applications.The IM injection success Test and Student Satisfaction and self-confidence scale were applied to the study and control groups after the laboratory application was completed.
  Arms: Working group

SUMMARY:
The study was conducted as a randomized controlled experimental study in order to determine the effect of hybrid simulation training on gaining the intramuscular injection skills of nursing students. The sample of the study consisted of 126 students (63 study groups, 63 control groups) enrolled in Nursing Principles Course at Pamukkale University Faculty of Health Sciences in 2018-2019 academic year. In the study, the study group performed hybrid simulation (standard patient+Digital half hip model simulator) and the control group performed simulation with low reality simulation method (hip/intramuscular model). Study data were collected using Student Identification Form, Intramuscular Injection Achievement Test, Intramuscular Injection Application Skill Assessment Form, Two Column Writing Reflective Thinking Strategies and Scale of Student Satisfaction and Self-confidence in Learning.

DETAILED DESCRIPTION:
Nursing students need to be proficient in nursing knowledge and skills before entering a health care environment in order to provide safe care to patients. One of the important and difficult to accomplish skills that nursing students must learn is the ability to administer intramuscular injections. In order to avoid complications due to IM injection application, it is necessary to comply with surgical asepsia, to know the method of application correctly and to have psychomotor skills. Therefore, nursing students are expected to graduate with knowledge and skills related to IM injection application during their education. Basic plastic mannequins without advanced technology, mannequins or models with low technological features that present the selected anatomical parts of the human body can also be used in standard patient and hybrid simulation. Hybrid simulation applications contribute to learners ' ability to develop psychomotor skills in a safe and realistic environment, as well as problem solving, critical thinking and decision making. Furthermore, hybrid simulations have become an ethical requirement to improve students ' skills without causing any potential harm to actual patients. In this study, the effectiveness of HS method will be evaluated to gain IM injection skills in nursing students. It will be ensured that the students ' knowledge and skills will be sufficient by increasing their desire to learn about IM injection, where they experience intense fear and anxiety before going to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Students who have not received IM injection skills training before,
* who have no clinical experience,
* who have accepted to participate in the research

Exclusion Criteria:

* Students who have received IM injection skills training before,
* who have clinical experience,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Intramuscular Injection Achievement Test | This test was administered 3 times. before the theoretical subject is explained, after the theoretical subject is explained and after the hybrid simulation is applied
  This test contains 21 multiple choice questions, including IM injection application topics.
Intramuscular Injection Application Skill Assessment Form | This test was administered 1 time. applied after hybrid simulation
  The IM injection application skill assessment form consists of 39 application steps. the total was calculated over 100 points.
Two Column Writing Reflective Thinking Strategies | This test was administered 1 time. applied after hybrid simulation
  In the case of two-column text used in this research, the page is divided horizontally in the middle. Two questions were asked on the left and right side of the page.
Scale of Student Satisfaction and Self-confidence in Learning | This test was administered 1 time. applied after hybrid simulation
  It consists of two sub-dimensions," satisfaction with learning "and" self-confidence", and a total of 13 items.

CONTACTS AND LOCATIONS:
Overall Officials: arife şanlıalp zeyrek, pHd, Principal Investigator — assistant researcher; nevin kuzu kurban, prof. dr, Study Director — responsible researcher
Locations (1):
- Turkey, Denizli, Pamukkale Universty Hospital, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study results will be announced in a publication
Supporting Information: Study Protocol
Time Frame: Findings can be shared after the study has been published.
Access Criteria: The sociodemographic characteristics of the participants, the test findings including the answers to the research questions and statistical analyzes will be shared.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

REFERENCES:
- [Background] Uys Y, Treadwell I. Using a simulated patient to transfer patient-centred skills from simulated practice to real patients in practice. Curationis. 2014;37(1):e1-e6. doi: 10.4102/curationis.v37i1.1184. Epub 2014 Nov 25. PMID 26852426